CLINICAL TRIAL: NCT03229239
Title: Implant the Corneal Stroma to the Diseased Cornea in Order to Cure Keratoconus
Brief Title: Corneal Stroma Implantation for the Treatment of Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170717
Record Dates: First submitted 2017-07-16; First posted 2017-07-25 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- corneal stroma implantation (Experimental): implant the corneal stroma to the diseased cornea of keratoconus patients
  Interventions: Procedure: corneal stroma implantation

INTERVENTIONS:
Procedure: corneal stroma implantation — During the operation,implant the corneal stroma to the diseased cornea of keratoconus.

SUMMARY:
The purpose of this study is to determine whether corneal stroma implantation is effective in the treatment of keratoconus.

DETAILED DESCRIPTION:
Keratoconus is a corneal disease with the progressive thinning of the central corneal stroma. The main treatment methods are corneal transplantation, corneal collagen cross-linking, etc. The effect of corneal collagen cross-linking is limited, and the lack of donor cornea is really a very big problem. In this pilot project, investigators would like to study whether corneal stroma implantation can increase the biomechanics of the cornea, which can, to some extent, delay the progress of keratoconus. This will allowed us to determine if useful data can be obtained, and if so, the donor cornea can be greatly saved.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced and completed keratoconus patients
2. Voluntarily signed informed consent
3. No surgery and anesthesia contraindications

Exclusion Criteria:

1. Acute edema of cornea
2. Primary keratoconus patients
3. The patients combined systemic diseases
4. Reject study and follow visit
5. Cannot tolerate surgery or anesthesia

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-08-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The best corrected visual acuity of the operated eye | 1 month after operation
  To check whether the best corrected visual acuity，which is scaled by the integrated refractometer,is improved after surgery.
The best corrected visual acuity of the operated eye | 3 months after operation
  To check whether the best corrected visual acuity，which is scaled by the integrated refractometer,is improved after surgery.
The best corrected visual acuity of the operated eye | 6 months after operation
  To check whether the best corrected visual acuity，which is scaled by the integrated refractometer,is improved after surgery.
The best corrected visual acuity of the operated eye | 12 months after operation
  To check whether the best corrected visual acuity，which is scaled by the integrated refractometer,is improved after surgery.

SECONDARY OUTCOMES:
The biomechanics of the operated eye | 1 month after operation
  To check whether the biomechanics,which is scaled by the corvis ST is improved after surgery.
The biomechanics of the operated eye | 3 months after operation
  To check whether the biomechanics,which is scaled by the corvis ST is improved after surgery.
The biomechanics of the operated eye | 6 months after operation
  To check whether the biomechanics,which is scaled by the corvis ST is improved after surgery.
The biomechanics of the operated eye | 12 months after operation
  To check whether the biomechanics,which is scaled by the corvis ST is improved after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Shi, sponsor, Study Chair — director of shandong eye hosiptal
Locations (1):
- Shandong Eye Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li N, Liu M, Tian G, Chen T, Lin Y, Qi X, Shi W, Gao H. Effects of femtosecond laser-assisted minimally invasive lamellar keratoplasty (FL-MILK) on mild-to-moderate and advanced keratoconus. Graefes Arch Clin Exp Ophthalmol. 2023 Oct;261(10):2873-2882. doi: 10.1007/s00417-023-06093-2. Epub 2023 May 12. PMID 37171602